CLINICAL TRIAL: NCT02952859
Title: Impact of Margin-accentuation IRE in Pancreatic Cancer
Acronym: IRE Marg
Status: Terminated | Type: Observational
Why Stopped: PI left hospital
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: IRE Marg
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Electroporation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- historic control group: Work-up and follow-up of the historic control will be performed through similar means by contacting primary care physicians and/or medical oncologists, if information cannot be received, the patient will be directly contacted. In case the patient cannot be reached and no other information can be received on patients outcome, the death registry will be contacted.
- comparator group: All patients with potentially and borderline resectable pancreatic cancer are potentially candidates for IRE and will be considered for this treatment. Patient will be recruited/referred through daily clinical practice from the Inselspital Bern. Final inclusion into the study will be performed by the responsible investigators at the Inselspital Bern. Patients will be included according to the inclusion/exclusion criteria mentioned.
  Interventions: Other: Irreversible electroporation

INTERVENTIONS:
Other: Irreversible electroporation
  Groups: comparator group

SUMMARY:
Pancreatic cancer is the fourth leading cause of cancer deaths overall and second after colon and rectum cancer among gastrointestinal cancers in Western countries. In Switzerland, 1,172 new pancreatic cancer patients were diagnosed in 2012. Unfortunately, only about 20% of pancreatic cancer patients present at a disease state that allows surgical resection while 30% have locally advanced, unresectable disease and 50% show distant metastases. While the latter two are currently treated in a palliative setting with median survival of at most 6-12 months, patients who undergo tumor resection with curative intentions also achieve only 5-year survival rates of 20-25% in best hands. The reasons for this poor outcome are thought to be chemoresistance, early establishment of metastatic disease, and importantly, high rates of R1 resections. Up to 80% of pancreatic resections have positive resection margins which are often found within the vascular groove and/or at the retroperitoneal margin, close to the superior mesenteric artery. This high rate of positive margins is only found after meticulous pathological work-up and is normally not detected after standard assessment of the specimen. However, the clinical importance of the high positivity of resection margin is even more highlighted as patients undergoing portal vein resection despite negativity of portal vein invasion after regular pathological work-up show significantly better survival compared to patients without portal vein resection. In sum, given the overall poor prognosis despite tumor resection, auxiliary treatment strategies to improve long-term outcomes are desperately needed. Over the last 5 years, irreversible electroporation (IRE) emerged as a non-thermal ablative modality that allows local tumor destruction with sparing vital structures like arteries, venous vessels, as well as the bile and pancreatic duct. There is increasing evidence that IRE for locally unresectable pancreatic cancer is effective with an increase in local progression free survival , distant progression free survival and overall survival compared to historic controls.Data on margin accentuation IRE are sparse while in a recent study published by Martin et al showed that margin accentuation among patients with borderline resectable disease can be performed safe and efficacious if the treatment can be performed "with a high degree of technical ability and skill set".

ELIGIBILITY:
Inclusion Criteria:

* Patients with histology proven or highly suspected potentially resectable or borderline resectable pancreatic cancer will be included.
* Age ≥ 18 years
* Able to undergo general anesthesia (ASA ≤ 3)
* Performance status ECOG <=2 (Eastern Cooperative Oncology Group)
* Life expectancy of at least 6 months
* Resectable or borderline resectable proven pancreatic adenocarcinoma of the pancreas

Exclusion Criteria:

* Cardiac conduction abnormalities (AV conduction abnormalities)
* History of epilepsy
* Recent history of myocardial infarction (2 months)
* Evidence of distant metastasis (e.g. liver, lung, peritoneum)
* Informed consent cannot be given by the patient
* Known hypersensitivity to the IRE electrodes (stainless steel 304L)
* Women of childbearing potential who are pregnant, breast feeding, or not taking an adequate method of contraception at the time of procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with potentially resectable and borderline resectable pancreatic cancer
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-01; Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Time from diagnosis to death for any reason | 6 weeks
  Postoperative complications
Time from diagnosis to death for any reason | 3 months
  Local and distal recurrence, cancer specific survival
Time from diagnosis to death for any reason | 6 months
  Local and distal recurrence, cancer specific survival
Time from diagnosis to death for any reason | 9 months
  Local and distal recurrence, cancer specific survival

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Worni, MD, Principal Investigator — Inselspital Berne
Locations (1):
- Inselhospital, Bern, Switzerland